CLINICAL TRIAL: NCT03614507
Title: Automation Oxygen Flow Titration in Spontaneously Breathing Infants Less Than One Year of Age During a First Episode of Bronchiolitis
Brief Title: Automation Oxygen Flow Titration in Spontaneously Breathing Infants
Acronym: FreeO2Bronchio
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: OXYNOV discontinues loan of FREEO2 devices
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FreeO2Bronchio (29BRC18.0091)
Record Dates: First submitted 2018-07-30; First posted 2018-08-03 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Bronchiolitis
Keywords: Hypoxemia; Infants; Oxygen therapy; Bronchiolitis
MeSH Terms: conditions — Bronchiolitis; Hypoxia

STUDY DESIGN:
Intervention Model Description: This is a multicenter, prospective, controlled, randomized, open-label study. Patients will be randomized to either the FreeO2 group for automatic oxygen titration or the manual group for oxygen therapy using manual flow titration.
Masking Description: The technology used does not allow blinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- FreeO2 group (Experimental): Automatic oxygen flow titration
  Interventions: Device: FreeO2 (modèle FO2-220-00) automatic oxygen flow titration
- Manual group (Active Comparator): Manual oxygen flow titration
  Interventions: Device: FreeO2 (modèle FO2-220-00) manual oxygen flow titration

INTERVENTIONS:
Device: FreeO2 (modèle FO2-220-00) automatic oxygen flow titration — Automatic adjustment of oxygen flow titration through the FreeO2 device. The monitor allows continuous monitoring and recording of SpO2 and Heart rate
  Arms: FreeO2 group
Device: FreeO2 (modèle FO2-220-00) manual oxygen flow titration — Manual oxygen flow titration performed by the healthcare provider in charge of the patient (nurse, physician). For this group, the FreeO2 device will only monitor and record SpO2 and heart rate.
  Arms: Manual group

SUMMARY:
The objective of this study is to assess the efficacy of the FreeO2 device in shortening the hospital length of stay during a first episode of hypoxemic bronchiolitis in infants less than 1 year of age.

FreeO2Bronchio study is a multicenter, prospective, controlled, randomized, open-label study.

DETAILED DESCRIPTION:
This is a controlled, randomized, open-label, multicentre trial. Patients will be included after written informed consent will be obtained from the patients' parents or legally authorized representatives. Patients will be randomized either in the "FreeO2" group for automatic oxygen flow titration or in the "manual" group for Oxygen therapy with manual flow titration. The SpO2 will be recorded continuously in both groups of the study using the FreeO2 device throughout the duration of hospitalization; In the group "FreeO2 ", the device will record the data continuously and allow the automation of oxygen titration - in the group "Manual", the device will only be used to monitor SpO2 and heart rate.

ELIGIBILITY:
Inclusion Criteria:

* Infants from 1 month of age and less than 1 year of age who present a first episode of bronchiolitis and require oxygen therapy
* Informed consent of parents (written informed consent will be obtained from the patients' parents or legally authorized representatives)
* Affiliation to the French social security system

Exclusion Criteria:

* Need for oxygen flow higher than 3 L / min to maintain SpO2 greater than 92%
* Patient with severity criteria according to the 2019 French National Authority for Health (HAS) guidelines and for whom it's indicated to maintain SpO2 above 94%
* Criteria of severity justifying from the start another technique of assisted ventilation:

  * Polypnea: respiratory rate (FR)> 80 c / min.
  * Consciousness with glasgow score (GSC) <or = 12. Hemodynamic instability (mean arterial pressure (MAP) <- 2 SD for age or use of vasopressors).
  * Cardiac or respiratory arrest.
  * PCO2> 55 mm Hg and pH <7.20 when blood gas are performed
* Need for urgent surgery
* Contraindication to the FreeO2 device as described in the user manual
* Lack of informed consent from parents
* Premature birth with a gestational age at birth under 36 weeks
* Severe co-morbidities (cystic fibrosis, immune deficiency, congenital heart disease, neuromuscular illness)

Ages: 1 Month to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 105 (Actual)
Dates: Start 2018-10-09 (Actual); Primary Completion 2023-07-05 (Actual); Study Completion 2023-07-05 (Actual)

PRIMARY OUTCOMES:
Length of hospital stay in hours since the admission to the emergency room. | 30 days max
  The length of hospital stay in hours since admission in the emergency room will be compared between the two groups.

SECONDARY OUTCOMES:
Number of patients readmited to hospital within 7 days and 30 days following discharge | 30 days max
Number of patients needing assisted ventilation (invasive or noninvasive ) | 30 days max
Number of patient admitted to the intensive care unit within 3 days following the hospital admission | 30 days max
Duration of enteral feeding (hours) | 30 days max
Duration of intravenous hydration (hours) | 30 days max
Number of reported Adverse Events | 30 days max
Time spent in the a area of severe desaturation (SpO2 <92%) and of hyperoxia area (SpO2> 98%). | 30 days max
Number of patients needing Heated Humidified High Flow Nasal Cannula (HFNNC) | 30 days max

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel ROUE, Dr, Principal Investigator — CHU de Brest
Locations (10):
- France (10):
  - La-Roche-Sur-Yon, Departmental Hospital Center, La Roche-sur-Yon, France
  - Limoges, University Hospital, Limoges, France
  - Lenval, University Hospital, Nice, France
  - Angers, University Hospital, Angers
  - Brest, University Hospital, Brest
  - CHI Créteil, Créteil
  - GHBS Lorient, Lorient
  - Marseille, University Hospital, Marseille
  - Nantes, University Hospital, Nantes
  - Rennes, university Hospital, Rennes

IPD SHARING:
Plan to Share IPD: No